CLINICAL TRIAL: NCT02225444
Title: A Prospective Study of Instrumented, Posterolateral Lumbar Fusions (PLF) With OsteoAMP® to Evaluate Long-Term Safety and Efficacy in Patients Requiring 1-2 Level Instrumented PLF
Brief Title: A Prospective Study of Instrumented, Posterolateral Lumbar Fusions (PLF) With OsteoAMP®
Status: Completed | Type: Observational
Sponsor: Bioventus LLC (Industry)
Collaborators: West Virginia University (Other); Rush University Medical Center (Other); University of Kansas (Other)
Responsible Party: Sponsor
Other Study IDs: TP1020
Record Dates: First submitted 2014-08-22; First posted 2014-08-26 (Estimated); Last update posted 2020-11-05 (Actual); Status verified 2020-11

CONDITIONS: Spondylolisthesis; Scoliosis; Intervertebral Disc Disease
Keywords: degenerative lumbosacral spine disease; posterolateral fusion evaluation; OsteoAMP; autograft
MeSH Terms: conditions — Spondylolisthesis; Scoliosis; Intervertebral disc disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- OsteoAMP treatment group: The OsteoAMP treatment group contains patients randomized to receive their own bone (retrieved from the surgical site) augmented with the OsteoAMP growth factor to assist with posterolateral arthrodesis at 1 or 2 adjacent levels between L1-S1.
  Interventions: Other: OsteoAMP

INTERVENTIONS:
Other: OsteoAMP — OsteoAMP in posterolateral fusion procedure of the lumbosacral spine

SUMMARY:
OsteoAMP is a novel allograft bone graft substitute (BGS) that has been processed to retain multiple endogenous growth factors for use in spinal fusion. The study is designed to obtain a higher level of clinical evidence for OsteoAMP in spinal fusion procedures and not to garner FDA regulatory approval. This is a prospective, non-randomized, non-controlled, multi-center study of OsteoAMP in instrumented, posterolateral lumbar fusion (PLF) in patients with degenerative disc disease, degenerative spondylolisthesis (up to grade 1), and/or mild degenerative scoliosis, up to 25 degree curvature. Patients that are scheduled to undergo instrumented, posterolateral spinal fusion surgery as part of their medical treatment and comply with the study eligibility criteria will be given the opportunity to consent and be entered into the study.

DETAILED DESCRIPTION:
The objective of this clinical study are: to evaluate the long term efficacy of OsteoAMP in patients requiring 1 to 2 adjacent level, instrumented posterolateral spinal fusion procedure of the lumbar or lumbosacral spine, and to evaluate OsteoAMP in spinal fusion procedures based on fusion results, adverse event rates, and pain and health scores.

Patients that are scheduled to undergo instrumented, posterolateral spinal fusion (PLF) surgery as part of their medical treatment and comply with the study eligibility criteria will be recruited and entered into the study. Subjects recruited into the study will receive OsteoAMP as part of an instrumented PLF surgical procedure. The surgery may also include nerve root decompressions through laminectomies and foraminotomies. As is consistent with the current standard of care.

The study involves consecutive patients suffering from lower back and leg pain due to degenerative disc disease (DDD), degenerative spondylolisthesis (up to grade 1), and/or mild degenerative scoliosis that are candidates for an instrumented PLF with pedicle screws in 1 or 2 motion segments of the lumbar or lumbosacral spine. Patients will require a total bone graft volume of at least 10cc per side per level in the PLF procedure, including OsteoAMP granules hydrated with bone marrow aspirate (BMA) and local autogenous bone.

Subjects will be followed for 24 months post-surgery.

ELIGIBILITY:
Summary of Inclusion Criteria:

1. Aged 21 to 85 years and skeletally mature at time of surgery
2. Diagnosis of degenerative disc disease (DDD), degenerative spondylolisthesis (up to grade 1), and/or mild degenerative scoliosis (up to 25°) curvature
3. One or more of the following are met: -instability (defined a angulation greater than or equal to 5 degrees and/or translation greater than or equal 4mm based on flexion/extension radiographs, -osteophyte formation, - decreased disc height, - thickening of ligamentous tissue, disc degeneration or herniation,- facet joint degeneration
4. Requires fusion (i.e., Symptomatic) at up to two contiguous levels from L1 to S1.
5. Preoperative ODI score of more than 30
6. Non-responsive to non-operative treatment for at least 6 months.
7. Lower back pain with or without claudication.
8. If of child-bearing potential, non-pregnant, non-nursing, and agrees to use contraception for up to 2 years following surgery
9. Willing and able to comply with study plan and able to understand and sign informed consent

Summary of Exclusion Criteria

1. Primary diagnosis of a spinal disorder other than DDD, degenerative spondylolisthesis up to Grade 1 or mild degenerative scoliosis of up to 25 degrees curvature
2. Requires fusion of more than 2 vertebral levels or of 2 non-adjacent vertebral levels
3. Conditions requiring medications that interfere with fusion or bone metabolism
4. More than one immobile vertebral level between L1 and S1 from any cause
5. Overt or active local or systemic infection, including latent infection around the surgical implantation site
6. Clinically severe obesity as defined by the National Institutes of Health
7. Uncontrolled diabetes mellitus as confirmed by HbA1c greater than 8%
8. History of osteoporosis or other metabolic bone disorders, including Paget's disease and osteomalacia
9. History of hypersensitivity to any of the agents used to process OsteoAMP
10. History of autoimmune disease
11. Received other bone graft substitutes
12. Received medication that may interfere with fusion or bone metabolism within 2 weeks of planned surgery
13. Received or plans to receive investigational therapy
14. Presence of active malignancy unless he/she has been treated with curative intent and there have been no clinical signs or symptoms of malignancy for at least 3 years
15. Presence of systemic disease or condition, which affects his/her ability to participate in the study requirements or the ability to evaluate the efficacy of the product
16. Prisoner, transient, or has been treated for chemical/alcohol dependency in an inpatient substance abuse program within 6 months prior to study enrollment or has significant psychosocial disturbance that would affect participation in the study, in the opinion of the investigator
17. Any condition for which the surgical procedure, in the opinion of the Investigator, poses an undue risk
18. Pursuing litigation related to cervical and/or lumbar/lumbosacral spine

Ages: 21 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male and female patients between 21 and 75 years old with degenerative disc disease, degenerative spondylolisthesis (up to grade 1), and/or mild degenerative scoliosis (up to 25° curvature) that have failed conservative treatment and are now indicated for instrumented posterolateral spinal fusion at 1 or 2 contiguous levels between L1-S1.
Sampling Method: Non-Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2015-11-19 (Actual); Primary Completion 2019-06-24 (Actual); Study Completion 2019-10-11 (Actual)

PRIMARY OUTCOMES:
Posterolateral fusion evaluation as determined by physician's assessment | 24 month follow up
  Radiographic evidence of fusion assessed by flexion-extension and CT radiograph or computed tomography (CT) scans.
  * Flexion extension radiographs timeframe: Pre-op, 6 month, 12 month, 24 months
  * CT timeframe: 12 month, 24 month. NOTE: If subject determined to be fused at 12 months, 24 month x-rays and CT not required
Improvement form baseline low back pain | 24 month follow up
  Improvement form baseline in low back pain and function as measured by Oswestry Disability Index (ODI)

SECONDARY OUTCOMES:
Improvements in pain | 24 month follow up
  Visual Analogue Scale (VAS) improvement from baseline to 24 month follow up assessed at timeframes: Pre-Op, 6 weeks, 3 month, 6 month, 12 month, 24 month
Improvements in function | 24 month follow up
  Short Form 36 (SF-36) score improvement compared to baseline at 24 months assessed at timeframes: Pre-Op, 6 weeks, 3 month, 6 month, 12 month, 24 month
Posterolateral fusion as determined by independently scored and adjudicated assessment | 24 month follow up
  Radiographic evidence of fusion assessed by flexion-extension and CT at 12 months and 24 months
Improvements in Other Health-Related Quality of Life measures | 24 month follow up
  Health-Related Quality of Life measures; work status, use of medication and perception of treatment effectiveness at Weeks 6 Post- Surgery, 3 months, 6 months, 12 months and 24 months

OTHER OUTCOMES:
Maintenance or improvement from baseline in neurological status with no new permanent deficits | 24 month follow up
  Neurological exam
Absence of serious product-related adverse events | 24 month follow up
  Serious product-related adverse events
Freedom from subsequent product-related surgical interventions | 24 month follow up
  Interventions include revision, removal, re-operation, and supplemental fixation at the affected level(s)

CONTACTS AND LOCATIONS:
Overall Officials: Scott Daffner, MD, Principal Investigator — West Virginia University; Howard An, MD, Principal Investigator — Rush University Medical Center
Locations (9):
- United States (9):
  - Yale University, New Haven, Connecticut
  - Rush University Medical Center, Chicago, Illinois
  - Kansas University Medical School, Kansas City, Kansas
  - Orthopedic Institute of Western KY, Paducah, Kentucky
  - William Beaumont, Royal Oak, Michigan
  - The Rothman Institute, Egg Harbor, New Jersey
  - OrthoCarolina Research Institute, Charlotte, North Carolina
  - St. Luke's University Health Network, Bethlehem, Pennsylvania
  - West Virginia University, Morgantown, West Virginia